CLINICAL TRIAL: NCT01250548
Title: The Controlled Trial of Apremilast for Rheumatoid Arthritis Treatment
Brief Title: The Controlled Trial of Apremilast for Rheumatoid Arthritis Treatment (CARAT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 009-293
Record Dates: First submitted 2010-08-26; First posted 2010-12-01 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; RA; Active rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Biological: apremilast
- Apremilast (Placebo Comparator): Placebo Compared to apremilast arm
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: apremilast — 30 mg BID apremilast taken orally for the first 12 weeks followed by responders randomized to either 30 mg BID apremilast (oral) or 30 mg BID placebo (oral) for 8 weeks
  Arms: 2
Other: Placebo
  Arms: Apremilast

SUMMARY:
The purpose of this study is to compare the effects of apremilast with a placebo (an inactive substance that looks like apremilast) on you and other people with rheumatoid arthritis.

The investigators will be collecting information in this study to help us determine -

* the safety of apremilast in patients with active rheumatoid arthritis
* how long it takes for patients with active rheumatoid arthritis to respond to apremilast
* how long the effects of apremilast last after the treatment has ended.

DETAILED DESCRIPTION:
Many manifestations associated with RA result from, or are significantly influenced by, the effects of pro-inflammatory cytokines (e.g., TNF, IL-1, IL-6). Specific inhibition of these cytokines with newer, parenterally administered biologic agents has revolutionized the treatment of RA. Apremilast is a novel, orally administered drug which approaches the reduction of pro-inflammatory cytokines via inhibition of phosphodiesterase type 4 (PDE4).

Apremilast, Acetamide, N-[2-[ (1S)-1-(3-ethoxy-4-methoxyphenyl)-2-(methylsulfonyl) ethyl]-2,3-dihydro-1,3-dioxo-1H-isoindol-4-yl] is a phosphodiesterase type 4 (PDE4) inhibitor under development for use in the treatment of inflammatory conditions.

PDE4 is one of the major phosphodiesterases expressed in leukocytes. Inhibitors of PDE4 cause accumulation of intracellular cyclic adenosine monophosphate (cAMP), which in turn activates protein kinase A and other downstream effectors, resulting in inhibition of pro-inflammatory cytokine transcription and other cellular responses such as neutrophil degranulation, chemotaxis, and adhesion to endothelial cells.

In human cellular models, apremilast inhibited production of inflammatory mediators such as TNF-α, IL-12, IL-2, IFN-γ, IL-5, IL-8, leukotriene B4 (LTB4), and the adhesion molecule CD18/CD11b (Mac-1).

Apremilast has also been shown to be a potent anti-inflammatory agent in several animal models of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to adhere to the study visit schedule and other protocol requirements
* documented rheumatoid arthritis (RA) diagnosis by the 1987 American College of Rheumatology (ACR) criteria for at least 6 months
* disease duration 6 or more months (from symptom onset)
* failed 1 or more DMARD
* active RA despite current DMARD therapy; active disease defined as 4 or more tender and 4 or more swollen joints (out of 28 joints examined) and any one of the following:
* ESR 28 or higher mm/hr;
* CRP 1.0 or more mg/dl;
* Morning stiffness 45 or more minutes.
* Patients receiving DMARD or biologic therapy must undergo a drug washout.
* Patients receiving a nonsteroidal anti-inflammatory drug (NSAID) and/or prednisone (10 or less mg day) must be on stable doses of these agents for more than 2 weeks.
* Must meet laboratory criteria as specified in the protocol
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening and must adhere to adequate forms of contraception as defined in the protocol. Must agree to pregnancy tests every 28 days while on study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication and for 28 days after taking the last dose of study medication

Exclusion Criteria:

* Inability to provide voluntary consent
* History of any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, neurologic, gastrointestinal, immunologic, or other major diseases
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or breastfeeding female
* Systemic fungal infection
* Active tuberculosis (TB) or a history of incompletely treated tuberculosis.
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
* Clinically significant abnormality on the chest x-ray (CXR) at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Use of any investigational medication within 28 days prior to randomization or 5 half-lives if known (whichever is longer)
* Any clinically significant abnormality on 12-lead ECG at screening
* History of congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID])
* History of Human Immunodeficiency Virus (HIV) infection
* Presence of hepatitis B surface antigens (HBsAg) or Hepatitis core antibody positive at screening.
* Antibodies to Hepatitis C virus at screening
* History of malignancy within 5 years prior to the screening visit (except for treated [i.e. cured] basal cell skin carcinomas and treated [i.e. cured] carcinoma in situ of the cervix)
* currently on DMARD therapy
* currently taking biologics
* treated with rituximab in the last 6 months
* Recent hospitalization (last 3 months)
* Planned pregnancy or major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine the time to response for subjects with active RA taking apremilast (30 mg per os [PO], twice per day [BID]) | 1.5 years

SECONDARY OUTCOMES:
Determine time to flare when apremilast is withdrawn | 1.5 years
Assess the efficacy and magnitude of response to apremilast in active RA measured by ACR 20, 50, & 70 response rates | 2 years
Assess safety of apremilast in subjects with active RA | 2 years
  Review of labs and possible adverse effects of study drug including Data Safety Monitoring Committee analysis.

CONTACTS AND LOCATIONS:
Overall Officials: John Cush, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor Research Institute - Arthritis Care and Research Center, Dallas, Texas, United States